CLINICAL TRIAL: NCT06843941
Title: The Effect of Music on Sleep Quality and Comfort Levels in Elderly Individuals: a Randomized Controlled Trial
Brief Title: The Effect of Music on Sleep Quality and Comfort in Elderly: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Derin Köksal, nurse, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 837; Decision No: 837 (Other: Izmir Bakırçay University Ethics Committee)
Record Dates: First submitted 2025-02-11; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Complementary and Alternative Therapies; Aging; Geriatric; Sleep Disorder in Elderly
Keywords: music theraphy; comfort; sleep quality; older adults
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Music Therapy; Complementary Therapies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Music Group (Experimental): For participants in the music group, the purpose of the study was explained before the music intervention, and after obtaining consent, the Individual Diagnosis Form, Richard-Campbell Sleep Scale, and Short Form General Comfort Scale were collected through face-to-face interviews. After the scales were completed, participants listened to the specially composed MusiCure® compositions via headphones and an mp3 player for 30 minutes each day over three days, between 19:00-21:00, considering non-intensive family visit hours and nursing care hours. After the music intervention, data were collected using the Richard-Campbell Sleep Scale and the Short Form General Comfort Scale on the morning of the fourth day after the third music session.
  Interventions: Other: Music intervention
- Control Group (No Intervention): For participants in the control group, the purpose of the study was explained, and after obtaining consent, the Individual Diagnosis Form, Richard-Campbell Sleep Scale, and Short Form General Comfort Scale were administered through face-to-face interviews. Data were collected again, without any intervention, on the morning of the fourth day using the Richard-Campbell Sleep Scale and the Short Form General Comfort Scale. No music intervention was provided to the control group. The control group will receive regular care and activities.

INTERVENTIONS:
Other: Music intervention — In the music group, "MusiCure®" compositions, which feature soft rhythmic melodies, were chosen. These musical pieces were composed by Danish composer Niels Eje (MusiCure, 2020) and are therapeutic in nature, designed for physical and mental relaxation within a range of 60-80 bpm (Eje, 2020). Literature reviews indicate that the "MusiCure®" album has positive effects on conditions such as pain, well-being, and anxiety (Fredriksson et al., 2009; Nilsson et al., 2009). The pieces to be used in this study were selected after communication with Niels Eje, and the recommended pieces were Winter, Early Spring, Equator, and Ocean Echoes (MusiCure, 2020). The music was presented hygienically to the participants through headphones and played for 30 minutes in four tracks via an mp3 player.
  Other Names: music; complemantary and alternative Therapies
  Arms: Music Group

SUMMARY:
The aim of this clinical study is to examine the effects of music on sleep quality and comfort levels in individuals aged 65 and older.

Background Sleep disorders in elderly individuals can negatively affect their comfort and quality of life. Due to its relaxing effect, music can be used as a supportive intervention in nursing care to improve sleep quality and comfort.

Methods

This study was conducted between January and April 2023 in the internal medicine department of a hospital in İzmir, Turkey. Patients aged 65 and older were divided into two groups using simple and stratified randomization:

Music group: Listened to MusiCure® compositions for 30 minutes, three times a week, for one week.

Control group: Received no intervention. Data Collection Process

Data were collected face-to-face on the first and fourth days. The following scales were used:

Richard Campbell Sleep Scale (to assess sleep quality) Short Form of the General Comfort Scale (to measure physical, psychological, and environmental comfort) Key Points Music intervention may positively affect sleep parameters such as sleep duration, sleep onset latency, and nighttime awakenings.

Music can increase psychological and physical relaxation, enhancing comfort levels in elderly individuals.

Considering individual music preferences may improve the effectiveness of the intervention.

Ethical Principles and Approvals The study was approved by the Clinical Research Ethics Committee of İzmir Bakırçay University and was conducted in accordance with the Helsinki Declaration.

This research aims to support the use of music interventions in nursing care and contribute to evidence-based practices to enhance sleep quality and comfort levels in elderly individuals.

DETAILED DESCRIPTION:
This study is a randomized controlled trial conducted to examine the effect of music intervention on sleep quality and comfort levels in individuals aged 65 and older.

Introduction and Background Sleep disorders in elderly individuals can negatively affect their quality of life and comfort levels. Non-pharmacological approaches stand out as alternative treatment methods due to their lack of side effects and cost-effectiveness. Music therapy is considered an important intervention for improving both sleep quality and overall comfort due to its relaxing effects.

Methods The study was conducted between January and April 2023 in the internal medicine department of a training and research hospital in İzmir, Turkey. Individuals aged 65 and older were included in the study. Participants were divided into two groups: the music intervention group and the control group.

Music group: Listened to MusiCure® compositions for 30 minutes, three times a week, for one week.

Control group: Received standard care without any intervention.

Data Collection Tools:

Richard Campbell Sleep Scale (to assess sleep quality) Short Form of the General Comfort Scale (to measure physical, psychological, and environmental comfort)

Randomization:

Patients were stratified by age (65-74, 75 and older) and gender and assigned to groups using a simple randomization method.

Key Points Music therapy may have positive effects on sleep quality parameters such as sleep duration, sleep onset latency, and nighttime awakenings.

Music can enhance psychological and physical relaxation, thereby increasing comfort levels in elderly individuals.

Considering individual music preferences may enhance the effectiveness of music interventions.

Ethical Principles and Approvals The study was approved by the Clinical Research Ethics Committee of İzmir Bakırçay University and was conducted in accordance with the Helsinki Declaration.

This research aims to provide a scientific basis for the use of music in nursing care and contribute to evidence-based practices to improve sleep quality and comfort in elderly individuals.

ELIGIBILITY:
Inclusion Criteria:

* (a) willingness to participate in the research, (b) proficiency in speaking and understanding Turkish, (c) being 65 years or older, (d) requiring hospitalization for at least one week.

Exclusion Criteria:

* (a) individuals with known hearing or visual impairments, (b) individuals with sleep disorders, (c) individuals diagnosed with advanced-stage diseases, (d) individuals with a history of cognitive disorders or a diagnosis of major depressive disorder.

Ages: 65 Days to 100 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Sleep Quality | Three days after the music intervention.
  This study aims to examine how music intervention affects the sleep quality of older individuals. Sleep quality was measured using the Richard Campbell Sleep Scale. This measurement evaluates various dimensions of sleep quality, including sleep duration, depth, frequency of awakenings, sleep onset latency, and environmental factors.

SECONDARY OUTCOMES:
Comfort Levels | Three days after the music intervention
  The general comfort levels of older individuals were measured using the Short Form of the General Comfort Scale. This measurement evaluates components of comfort, including physical ease, emotional comfort, environmental comfort, and social comfort.

CONTACTS AND LOCATIONS:
Overall Officials: yasemin yıldırım, prof.dr., Study Director — Ege University Faculty of Nursing
Locations (1):
- Buca Seyfi Demirsoy Training and Research Hospital, Izmir, buca, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All data will be stored for at least 15 years after the completion of the study. All personal and medical information of the participants will remain confidential. Even in the case of publication of the research results, the identity of the individuals will remain anonymous

REFERENCES:
- [Background] Music Therapy. (2020). Applications-Extended information about music research and practice. MusiCure.
- [Background] Eje, I. (2020). MusiCure®: A therapeutic music selection developed to promote physical and mental relaxation in hospital environments, using a 60-80 bpm range. Retrieved from https://www.musicurestream.com
- [Background] Ziv N, Rotem T, Arnon Z, Haimov I. The effect of music relaxation versus progressive muscular relaxation on insomnia in older people and their relationship to personality traits. J Music Ther. 2008 Fall;45(3):360-80. doi: 10.1093/jmt/45.3.360. PMID 18959456
- [Background] Richards K. Techniques for measurement of sleep in critical care. Focus Crit Care. 1987 Aug;14(4):34-40. No abstract available. PMID 3650169
- [Background] Fredriksson AC, Hellstrom L, Nilsson U. Patients' perception of music versus ordinary sound in a postanaesthesia care unit: a randomised crossover trial. Intensive Crit Care Nurs. 2009 Aug;25(4):208-13. doi: 10.1016/j.iccn.2009.04.002. Epub 2009 May 14. PMID 19446459
- See also: It was used for simple and stratified randomization — https://www.randomizer.org